CLINICAL TRIAL: NCT04589221
Title: Sensory and Oral Processing Characteristics of Commonly Consumed Foods
Status: Completed | Type: Observational
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, Vicki Tan, Senior Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Other Study IDs: 2019-084
Record Dates: First submitted 2020-10-07; First posted 2020-10-19 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Adults
Keywords: Eating behaviour; Eating rate; Texture; Sensory
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Degree of food processing and food texture: Processed vs unprocessed foods based on NOVA classification
  Soft and hard foods manipulated by cooking method
  Interventions: Behavioral: Ad libitum energy intake

INTERVENTIONS:
Behavioral: Ad libitum energy intake — Investigate ad libitum energy intake according to degree of food processing and eating behaviour

SUMMARY:
Rationale: Oral processing behaviours (i.e. eating rate, bite size, chews per bite) play an important role in the onset of satiation and satiety and laboratory studies have shown that people who eat quickly consume more energy during an ad libitum meal. Therefore, one possible approach to control the energy intake is to encourage eating behaviour that slow the rate of calorie intake of the meal. Numerous studies that use external cues and prompts to change the eating rate (e.g. utensil, devices) have shown to produce clinically meaningful results. However, the long-term efficacy of these external manipulation to eating rate remains unclear and have difficulties in adherence. Texture led changes to oral processing behaviours therefore offer an exciting opportunity to adapt an individual's response to structure properties of the food being consumed in a way that maintains the associated eating experience and satiety from food intake.

However, no studies to date have investigated how differences food processing influence food texture characteristics and oral processing behaviour and the subsequent impact on energy intake for commonly consumed meals. The proposed study will explore the impact of food texture and oral processing characteristics on energy intake for the minimally-processed and ultra-processed foods or meals, to explore the impact of food processing on texture, oral processing and energy intakes.

Objective: The objectives of the study are to characterise the differences in sensory perception, and oral processing behaviours (i.e. eating rate, bite size, chew per bite, oral exposure time etc.) of foods and meals that differ in their degree of processing (Part 1), and to further investigate how texture-based differences in oral processing behaviour influence ad-libitum energy intake (Part 2). This study is also aimed to see how is the texture-based differences in oral processing behaviour modified by degree of food processing (i.e. un-, minimally-processed, processed and ultra-processed foods) (Part 2).

Study design: Part 1) Randomised non-blinded feeding trial where participants taste up to 48 food items over 3 test sessions; Part 2) 2x2 randomised crossover design where participants receive 4 treatments (i.e. 4 test meals) over 4 test sessions

Study population: Healthy females and males (n=30 for Part 1; n=50 for Part 2) aged 21-50 years with BMI between 18-25 kg/m2

Intervention: Part 1) Participants will taste and evaluate up to 48 food items over 3 sessions in randomised order. Session 1 involves tasting of up to 16 food items and computer task to rate and evaluate their perception and health behaviour. Sessions 2-4 involve evaluation of sensory characteristics, video-recordings of participants eating, and wrist worn accelerometer to track wrist movement while tasting up to 48 food items.

DETAILED DESCRIPTION:
Objectives:

The objectives of the study are to characterise the differences in sensory perception, and oral processing behaviours (i.e. eating rate, bite size, chew per bite, oral exposure time etc.) of foods and meals that differ in their degree of processing, and to further investigate how texture-based differences in oral processing behaviour influence ad-libitum energy intake. In addition, this study is also aimed to see how is the texture-based differences in oral processing behaviour modified by degree of food processing (i.e. un-, minimally-processed, processed and ultra-processed foods).

Study Design:

The study involves 2 parts. A maximum of 30 participants will be recruited to complete Part 1 (1 screening session & 3 test sessions); and a maximum of 50 participants will be recruited to completed Part 2 (4 test sessions) of the study.

Part 1) Sensory perception and health behaviour for foods varying in degree of processing and nutrient source will be evaluated using a Health Behaviour Questionnaire and food perception and health behaviour task. Perceived sensory and oral processing behaviour differences between a series of commercially available and commonly consumed foods (e.g. carrot, apple, meatball, etc.) will be assessed using sensory descriptive analysis on 100mm Visual Analogue Scale (VAS), and video recording, respectively.

Part 2) In addition, the sensory and oral processing behaviour, satiety and ad-libitum energy intake across different meals (e.g. rice with meat and vegetable, meat with potato and salad, etc.) will be assessed using video recording, sensory and appetite assessment on 100mm VAS, and a weighing food balance.

The current study will require participants to attend either 4.5 hours (Screening and Part 1), 9.5 hours (Screening and Part 2) or 12.5 hours (Screening, Parts 1 and 2). All participants will be required to join for one-time screening prior to the study. Participants will require to fast for three-hour (Part 1) and at least one hour (Part 2) before their scheduled lunch-time test sessions. Each session will last for approximately one hour (Screening, Part 1), or two hours (Part 2), as indicated accordingly.

In the situation of participant dropout, the data that have been collected until the time of withdrawal will be kept and analysed. The reason is to enable a complete and comprehensive evaluation of the study.

Test Foods:

Part 1) Commercially available and commonly consumed foods (e.g. carrot, apple, meatball, etc.) Part 2) Consist of components previously tested in Part 1 and comprise foods that are commercially available, safe for human consumption and prepared in line with safe hygienic food preparation (e.g. rice with meat and vegetable, meat with potato and salad, etc.)

Screening (Session 1, 1- 1.5 hour):

All potential participants will be asked to give informed consent before taking part in any of the research activities. Participants are to complete a screening questionnaire and to taste five different basic taste solutions (sweet [sucrose, 3.2-100 mmol/L], salty [sodium chloride, 3.2-100 mmol/L], bitter [caffeine, 0.25-0.79 mmol/L], sour [citric acid, 0.63-5 mmol/L] and umami[monosodium glutamate, 1-31.6 mmol/L]) to assess their taste discrimination ability. Basic anthropometric measurements such as height, weight, skinfold measurements and percentage body fat using a Bioelectrical Impedance Analyser will be taken.

Successfully screened participants will proceed to complete a Health Behaviour Questionnaire and taste no more than 16 samples to rate and evaluate their perception and health behaviour for the foods varying in degree of processing and nutrient sources at the remaining of the screening session.

Part 1 (3 test sessions, 1 hour each):

Sensory and oral processing behaviour of commercially available food samples will be assessed. A maximum of 30 participants will be recruited for this part of the study. Participants will taste no more than 16 samples in each session.

Participants will be asked to taste each food sample and evaluate on liking, familiarity and the sensory attributes such as overall flavour intensity, firmness, crunchiness, chewiness, saltiness and sweetness. A mandatory inter-stimulus break of one minute will be enforced between each sample to reduce possible fatigue and allow time to cleanse your palate with water and crackers provided. All evaluations will be administrated and collected using a computer. Participants will also be video-recorded during the sessions for collection of oral processing data (i.e. eating rate, bite number, bite size etc). In addition, Participants will be asked to wear a wrist worn accelerometer (M5StickC ESP32-PICO Mini loT Development Kit, China) on the hand they eat with to track the wrist movement while eating.

Part 2 (4 test sessions, 2 hour each):

The sensory, oral processing characteristics and ad libitum energy intake for different meals will be assessed in this part. A maximum of 50 participants will be recruited for this part of the study. Participants who completed Part 1 will be invited to join the Part 2, however the participation is not mandatory. Participants will attend 1 session per week for four consecutive weeks to evaluate up to 4 ad libitum test meal across for lunch-time sessions, i.e. 1 ad libitum test meal per session.

Participant will be required to fast from 11.00 pm the evening before and refrain from engaging in vigorous physical activities.

On each test day, participants will be asked to arrive at CNRC between 8.00-9.00am and complete a set of appetite ratings disguised as "Mood Questions" (pre-breakfast rating). Following the pre-breakfast rating, participants will receive a standardised, fixed portion breakfast and mid-morning drink/snack to take away with them and consume at fixed intervals during the morning (before the lunch). The purpose is to equilibrate their appetite need state ahead of the ad-libitum test meal at lunch session.

Participants will consume the breakfast within 15 minutes, after which complete a second set of appetite ratings (post-breakfast ratings). Participants will refrain from consuming anything except water and continue to complete the appetite rating at 15 or 30 minutes' intervals, prompted with reminder set on their mobile device.

After approximately 2 hours, participants will consume the mid-morning drink/ snack within 15 minutes. Participants will then continue to rate their appetite at 15 minute intervals before coming to CNRC for their lunch.

The lunch session will be scheduled from midday onwards and will begin with a set of appetite rating (pre-lunch rating). Participants will be served an ad libitum test meal (~800g to 1000g) along with a glass of water, and instructed to taste a mouthful of the meal and rate its sensory characteristics. Participants will then be asked to consume the ad libitum test meal in their normal way and to eat until comfortably full. Participants' eating behaviour at lunch will be recorded in order to analyse and behaviourally code their oral processing behaviour (i.e. eating rate, bite number, bite size etc). In addition, Participants will be asked to wear a wrist worn accelerometer on the hand they eat with to track the wrist movement while eating. After completed eating, participants will be required to complete post-lunch appetite ratings at 15minutes interval for 90minutes, and bring a food diary home for recording their food and beverage intake for the rest of the test day.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female
* Aged between 21 and 50-year-old
* Are of normal weight (BMI 18-25kg/m2)
* Stable weight for the previous 12 months (<5kg weight fluctuation in the previous year)
* Healthy dentition and ability to bite, chew and swallow normally
* No history of pain or discomfort in jaw movements or excessive teeth clenching or grinding
* No caries or periodontal disease

Exclusion Criteria:

* Smoker
* Currently pregnant or in lactating
* Dislikes, intolerances or allergies to foods or common food ingredients e.g. nuts, soya, wheat, gluten, cereal, fruits, biscuits, dairy products, rice, vegetable, meat, seafood, sugar and sweetener, gelatin, natural food colouring or flavourings (e.g. MSG), etc.
* Have any specific dietary requirements and/ or restrictions (e.g. Vegan/ vegetarian, religious beliefs, lactose intolerance, calorie restricted diet etc.)
* Sinus problems that affect your taste and smell
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Taking insulin or medication known to affect your appetite or metabolism
* Have major chronic diseases such as heart disease, cancer or diabetes mellitus
* Have active Tuberculosis (TB) or currently receiving treatment for TB
* Have any known Chronic Infection or known to suffer from or have previously suffered from or is a carrier of Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), Human Immunodeficiency Virus (HIV)
* Member of the research team or their immediate family members. Immediate family member is defined as a spouse, parent, child, or sibling, whether biological or legally adopted
* Enrolled in a concurrent research study judged not to be scientifically or medically compatible with the study of the CNRC

Ages: 21 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: General public of Singapore aged between 21 to 50 years old.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Oral processing behaviour | Part 1, during the 3 test sessions, up to 1 hour each
  Participants will be video-recorded to measure oral processing behaviour of the test foods
Ad libitum energy intake | Part 2, during the 4 test sessions, up to 2 hours each
  Test foods consumed during test sessions by the participants will be recorded.
  Participants will be asked to bring a food dairy home for recording their food and beverage intake for the rest of the test day.

CONTACTS AND LOCATIONS:
Overall Officials: Pey Sze Teo, PhD, Principal Investigator — Teo_Pey_Sze@sifbi.a-star.edu.sg
Locations (1):
- Singapore Institute of Food and Biotechnology Innovation (SIFBI)/Clinical Nutrition Research Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Teo PS, Lim AJ, Goh AT, R J, Choy JYM, McCrickerd K, Forde CG. Texture-based differences in eating rate influence energy intake for minimally processed and ultra-processed meals. Am J Clin Nutr. 2022 Jul 6;116(1):244-254. doi: 10.1093/ajcn/nqac068. PMID 35285882